CLINICAL TRIAL: NCT00362024
Title: MK0952 in Patients With Mild-to-Moderate Alzheimer's Disease
Brief Title: MK0952 in Patients With Mild-to-Moderate Alzheimer's Disease (0952-004)(COMPLETED)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0952-004; 2006_026
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — MK-0952

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0952
Drug: Comparator: Placebo

SUMMARY:
MK0952 is a phosphodiesterase type IV (PDE4) inhibitor in development for improvement of cognitive impairment in mild-to-moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or females
* Age >/= 55 years, With mild-to-moderate AD, with MMSE between 18 and 26, inclusive, MHIS score </= 4, Global CDR score of 1 or 2
* Who have a reliable informant/caregiver to accompany patient to all clinic visits
* If using a symptomatic AD treatments, patients must be on stable dose for >/= 6 months

Exclusion Criteria:

* Patients must not be living in nursing home or skilled nursing facility
* Patients must not have current evidence and/or history of Crohn's disease, ulcerative colitis, proctitis, GI bleeding, mesenteric arteritis
* Patients must not have current evidence and/or history of poorly-controlled hypertension, clinically significant cardiac arrhythmia, angina, or CHF
* Patients must not have current evidence and/or history of a psychotic disorder or major untreated depressive disorder
* Patients must not have current evidence and/or history of stroke or multiple lacunar infarcts, or neurological or neurodegenerative disorder (other than AD)
* Various concomitant therapy restrictions

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC